CLINICAL TRIAL: NCT06044025
Title: A Feasibility Study Evaluating a Role for Maintenance Therapy in Patients With Biochemically Progressive Castration Sensitive Prostate Cancer on Intermittent Androgen Deprivation Therapy
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 274850
Record Dates: First submitted 2023-08-29; First posted 2023-09-21 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Castration Sensitive Prostate Cancer
MeSH Terms: interventions — Metformin; Curcumin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Metformin + Turmeric (Experimental): Each subject will begin using metformin and turmeric within 7 days of consent. Subjects will start with metformin 500 mg by mouth (po) two times daily (bid) with meals for 14 days. Metformin titration will then increase to 850 milligram (mg) po bid for 14 days before increasing titration to a desired dosage of 1,000 mg po bid. For those subjects currently taking Metformin, they will continue current dose (if 1,000 mg po bid) or titrate dose as just described until maximum dose is achieved.
  After two weeks of metformin titration, each subject will start with 1,500 mg turmeric po daily with meals. Dose can be temporarily reduced to 1,000 mg po daily for those who report GI discomfort. If GI discomfort has resolved within one month of the dose reduction, subjects will resume 1,500 mg po daily. If GI discomfort has not resolved the participant may be insturcted to stop taking the study treatment and be removed from the study.
  Interventions: Drug: Metformin; Drug: Turmeric

INTERVENTIONS:
Drug: Metformin — Subjects will start with metformin 500 mg by mouth (po) two times daily (bid) with meals for 14 days. Metformin titration will then increase to 850 milligram (mg) po bid for 14 days before increasing titration to a desired dosage of 1,000 mg po bid. For those subjects currently taking Metformin, they will continue current dose (if 1,000 mg po bid) or titrate dose as just described until maximum dose is achieved.
Drug: Turmeric — Each subject will start with 1,500 mg turmeric po daily with meals. The dose can be temporarily reduced to 1,000 mg po daily for those who report GI discomfort. If GI discomfort has resolved within one month of the dose reduction, subjects will resume 1,500 mg po daily. If GI discomfort has not resolved or resumes at increased dose, the subject may be instructed to stop taking the study treatment and removed from the study.

SUMMARY:
The goal of this clinical trial is to assess the feasibility of adding a combination of metformin and turmeric as part of a nutritional intervention regimen to the current standard of care, namely, intermittent Androgen Deprivation Therapy (iADT), for patients with castration sensitive biochemical progressive prostate cancer.

The main objectives are:

* Assess the feasibility of the study population and enrollment.
* Evaluate time to PSA relapse with nutritional intervention on iADT.

Participants who are receiving iADT will be dispensed Metformin and turmeric and complete a pill diary. Participants will also have blood and stool samples collected and complete quality of life questionnaires.

The long-term goal is to further assess the efficacy and safety of this nutritional regimen and the roles of metabolic syndrome, microenvironment/microbiome, and genomic vs epigenomic profiles in the care of these patients through a clinical trial.

DETAILED DESCRIPTION:
The purpose of this research is to determine if a nutritional plan of metformin and turmeric is feasible for individuals receiving iADT for prostate cancer. Turmeric is an over-the-counter supplement that is believed to provide anti-inflammatory effects. Metformin is an FDA-approved medication for diabetes to help lower blood sugar. This feasibility study will be conducted according to the standard of care (SoC) for eligible subjects receiving iADT but coordinated and streamlined in a prospective manner to care for subjects while collecting and annotating data for the duration of their care.

All subjects will receive iADT + turmeric + metformin + dietary consultation.

SoC laboratory tests will be performed in accordance with clinical practice for the care of patients with prostate cancer on or off iADT. Additional vials of blood will be collected for research purposes in order to assess epigenetic biomarkers, CSC biomarkers, and cancer dormancy biomarkers. Stool samples will be used to obtain microbiome profiles. QOL instruments (FACT-P and AMS) will also be administered.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older.
* History of prior prostatectomy and/or radiation therapy to the prostate.
* Currently have rising PSA levels ≥ 0.2 ng/ml if they have undergone radical prostatectomy, or a PSA ≥ nadir + 2 if they have received only radiotherapy. Patients who were not offered salvage radiotherapy as an alternative treatment will be considered ineligible (due to a high PSA, other medical concerns).
* Currently have at least 2 consecutively rising serum PSA levels more than 1 week apart
* Currently have a PSA doubling time < 9 months obtained within 60 days of consent.
* Eugonad with testosterone > 150 ng/dl at time of consent.
* Prior ADT (including iADT) for up to 24 months in association with definitive treatment is permitted if completed at least 12 months prior to consent.
* Eastern Cooperative Oncology Group (ECOG) performance status 0 - 1.
* Willing to take study agents at the dose specified with meals.
* Willing to discontinue current vitamin/mineral supplements and use only those provided by study. Herbal supplements may still be used.

Exclusion Criteria:

* Current Chronic Lymphocytic Leukemia (CLL), Monoclonal Gammopathy of Unknown Significance (MGUS), Renal Cell Carcinoma (RCC) or another cancer requiring active treatment. Indolent or stable malignancies such as non-melanoma skin cancers are allowed.
* Any active or deteriorating liver or renal disease, Human Immunodeficiency Virus (HIV), Hepatitis B, Hepatitis C or bone marrow deficiency.
* Any history of allergic reactions attributed to turmeric, metformin, or other compounds of similar chemical or biologic compositions.
* History of lactic acidosis or risk factors for lactic acidosis (e.g., renal impairment, concomitant use of carbonic anhydrase inhibitors such as topiramate, hypoxic states such as acute congestive heart failure, excessive alcohol intake, and hepatic impairment).
* Any other condition that, in the opinion of the investigator, might interfere with the safe conduct of the study.

Ages: 18 Years to 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2024-04-11 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
Assess feasibility of recruitment | 12 months of enrollment being open
  Assessed using frequency (in percentage) of the number of subjects enrolled in the first six and twelve months out of the total desired accrual
Evaluate time to PSA relapse with nutritional intervention on iADT. | up to 27 months
  Observed from the time of consent to the time of PSA relapse or at the end of the study period (i.e., 27 months), whichever comes first. A survival curve will be used to estimate the accumulated rate of PSA relapse over time (over 27 months).

SECONDARY OUTCOMES:
Quality of life (QOL) assessed by the Functional Assessment of Cancer Therapy-Prostate (FACT-P), Version 4. | up to 27 months
  Obtain Functional Assessment of Cancer Therapy-Prostate (FACT-P) scores at baseline, after completion of 8 months of iADT with nutritional intervention, and at the end of the study (i.e., after 27 months). Minimum and maximum values 0-156. Higher scores indicate better outcome.
Quality of Life (QOL) assessed by the Aging Male Symptoms Questionnaire (AMS Questionnaire). | up to 27 months
  Obtain Aging Male Symptoms Questionnaire (AMS Questionnaire) scores at baseline, after completion of 8 months of iADT with nutritional intervention, and at the end of the study (i.e., after 27 months). Minimum and maximum values 17-85. Higher scores indicate worse outcome.

OTHER OUTCOMES:
Expression levels of Metabolomic biomarkers from blood samples | up to 16 months
  Assessed at baseline, after 8 months of iADT with nutritional intervention, and at 16 months, and will be summarized using mean ± standard deviation and/or median (min, max)
Expression levels of CSC biomarkers including EMT and miRNAS from blood samples | up to 16 months
  Assessed at baseline, after 8 months of iADT with nutritional intervention, and at 16 months, and will be summarized using mean ± standard deviation and/or median (min, max)
Expression levels of Cancer dormancy Biomarkers (miR-200s, TGF-beta, BMPs, immune and inflammatory factors) from blood samples | up to 16 months
  Assessed at baseline, after 8 months of iADT with nutritional intervention, and at 16 months, and will be summarized using mean ± standard deviation and/or median (min, max)
Microbiome profiling from the stool samples to assess gut microbiome | up to 16 months
  Assessed at baseline, after 8 months of iADT with nutritional intervention, and at 16 months, and will be summarized using mean ± standard deviation and/or median (min, max)

CONTACTS AND LOCATIONS:
Overall Officials: Shi-Ming Tu, MD, Principal Investigator — University of Arkansas
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States